CLINICAL TRIAL: NCT05631951
Title: Bone Transport Through Induced Membrane Technique Versus Conventional Bone Transport Technique in Management of Bone Defects of Lower Limbs
Brief Title: Bone Transport Through Induced Membrane vs Conventional Bone Transport in Management of Bone Defects of Lower Limbs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD57/2020
Record Dates: First submitted 2022-11-01; First posted 2022-11-30 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: 30 patients were included and divided randomly into two equal groups:
  * Group (A) will undergo BTM
  * Group (B) will undergo BT
  Methods:
  I. Preoperative evaluation
  II. Operative interventions:
  A. Pre-operative:
  B. Operative interventions
  * first step
    • resection of infected bone
  * Second step:
  (A) Group A cement spacer and external fixator were applied then removal of cement spacer and metaphyseal osteotomy done (B)Group B
  * external fixator was applied then metaphyseal osteotomy done C. Post-operative
  * bone transport was started after latency of 7 days (from osteotomy) at rate of 1mm per day in 4 increments per day (rhythm of 0.25 mm every 6 hours) until reaching docking site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bone transport through induced membrane (Active Comparator): First stage
  1. antibiotic impregnated cement spacer was applied to the bone defect
  2. external fixator was applied for 6-8 weeks ϖ Second stage
  1.removal of cement spacer done 2.metaphyseal osteotomy done
  Interventions: Procedure: bone transport through induced membrane
- bone transport (Active Comparator): 1. removal of all hardware
  2. resection of infected bone segments
  3. external fixator was applied
  4. metaphyseal osteotomy done
  Interventions: Procedure: bone transport

INTERVENTIONS:
Procedure: bone transport through induced membrane — Debridement done followed by external fixator and cement application to be followed by removal of cement (after 6 weeks) and start bone transport
  Arms: bone transport through induced membrane
Procedure: bone transport — Debridement done then external fixator was applied then bone transport started.
  Arms: bone transport

SUMMARY:
This is a prospective randomised controlled comparative study comparing bone transport through induced membrane (BTM) and conventional bone transport (BT) in management of bone defects in infected non united fractures of long bones of lower limbs (femur, tibia) as regard clinical, functional outcomes and possible complications.

DETAILED DESCRIPTION:
A prospective randomised controlled study was conducted at Ain shams university hospitals. A total of 30 patients with infected non united fractures of long bones of lower limbs (femur and tibia) were divided randomly into 15 patients treated by bone transport through induced membrane technique (BTM) (Group A) and 15 patients treated by conventional bone transport technique (BT) (Group B)

ELIGIBILITY:
Inclusion Criteria:

* Sex: both sexes.
* Age:18-60 yrs old.
* Lesion: tibial or femoral bone defects (>4 cm)
* Defects resulting from infected non-united fractures

Exclusion Criteria:

* Pathological and congenital defects
* Aseptic traumatic bone defects
* Defects less than 4 cm
* Multiple defects Pediatric age group

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
External fixation time | through study completion, an average of 1 year
  time from the initial application of the fixator until removal of fixator (in months)
External fixation index | through study completion, an average of 1 year
  calculated by dividing the EFT (months) by the bone defect size (centimeters)
Docking time | through study completion, an average of 1 year
  time taken (months) from end of bone transport till union of docking site (both with and without bone graft)
Association for the Study and Application of the Method of Ilizarov (ASAMI) Scoring System | through study completion, an average of 1 year
  scoring system for bone and functional results
complications rate | through study completion, an average of 1 year
  number of complications in each group
additional operations | through study completion, an average of 1 year
  number of additional operations in each group

CONTACTS AND LOCATIONS:
Overall Officials: Mootaz F Thakeb, MD, Study Chair — Professor Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marais LC, Ferreira N. Bone transport through an induced membrane in the management of tibial bone defects resulting from chronic osteomyelitis. Strategies Trauma Limb Reconstr. 2015 Apr;10(1):27-33. doi: 10.1007/s11751-015-0221-7. Epub 2015 Apr 4. PMID 25840909
- [Background] Uzel AP, Lemonne F, Casoli V. Tibial segmental bone defect reconstruction by Ilizarov type bone transport in an induced membrane. Orthop Traumatol Surg Res. 2010 Apr;96(2):194-8. doi: 10.1016/j.rcot.2010.02.001. PMID 20417920